CLINICAL TRIAL: NCT00000219
Title: Buprenorphine Dose Alteration Study
Brief Title: Buprenorphine Dose Alteration Study - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-06969-1; R18DA006969 (NIH); R01-06969-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 1992-04

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to examine the effects in buprenorphine dose alterations in opioid dependent individuals being maintained on buprenorphine.

ELIGIBILITY:
Please contact site for information.

Ages: 19 Years to 41 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1991-12; Study Completion 2001-07

PRIMARY OUTCOMES:
Opioid withdrawal
Subjective dose estimate
Drug effect characteristics: ARCI
Physiological changes in: pupil diameter
Physiological changes in: blood pressure
Physiological changes in: heart rate
Physiological changes in: respiration
Physiological changes in: skin temperature

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States

REFERENCES:
- [Background] In preparation. In preparation.